CLINICAL TRIAL: NCT01377376
Title: A Phase 3, Randomized, Double-Blinded, Placebo-Controlled Study of ARQ 197 Plus Erlotinib Versus Placebo Plus Erlotinib in Previously Treated Subjects With Locally Advanced or Metastatic, Non-Squamous, Non-Small-Cell Lung Cancer With Wild-type Epidermal Growth Factor Receptor
Brief Title: A Phase 3, Randomized, Double-Blinded, Placebo-Controlled Study of ARQ 197 Plus Erlotinib Versus Placebo Plus Erlotinib
Acronym: ATTENTION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARQ197-006
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ARQ 197; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ARQ 197 (Experimental): ARQ 197 and Erlotinib
  Interventions: Drug: ARQ 197 and Erlotinib
- Placebo (Placebo Comparator): Placebo and Erlotinib
  Interventions: Drug: Placebo and Erlotinib

INTERVENTIONS:
Drug: ARQ 197 and Erlotinib — Oral twice daily administration of ARQ197 and oral once daily administration of erlotinib
  Arms: ARQ 197
Drug: Placebo and Erlotinib — Oral twice daily administration of placebo and oral once daily administration of erlotinib
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine if the combination regimen of ARQ 197 with erlotinib will improve overall survival (OS) compared to erlotinib monotherapy in subjects with locally advanced or metastatic non-squamous NSCLC with wild-type EGFR who have received 1 or 2 prior systemic anti-cancer therapies in the Intent-to-Treat (ITT) population.

ELIGIBILITY:
Inclusion Criteria

1. Male or female at least 20 years of age with life expectancy ≥ 3 months
2. Histologically or cytologically confirmed surgically unresectable locally advanced or metastatic (stage IIIB/IV) non-squamous NSCLC with wild-type (excluding major activating mutation (exon 19 deletion and/or exon 21 L858R mutation)) EGFR gene status confirmed by a highly sensitive PCR assay
3. Evaluable disease according to RECIST, Version 1.1
4. Received one or two prior lines of systemic anti-cancer therapy for advanced or metastatic disease, one of which must be a platinum-based therapy
5. ECOG performance status of 0 or 1
6. Demonstrate adequate bone marrow, liver, and renal functions, defined as:

   • ALT and AST ≤ 2.5 × upper limit of normal (ULN), total bilirubin ≤ 1.5 × ULN, ANC ≥1.5 × 10^9/L, platelet count ≥100 × 10^9/L, hemoglobin ≥9.0 g/dL, and serum creatinine ≤1.5 mg/dL.
7. Voluntary written informed consent form before performance of any study-specific procedures or tests

Exclusion Criteria

1. Prior therapy with an EGFR inhibitor and/or tivantinib
2. Any systemic anti-tumor treatment for NSCLC or investigational agents within 4 weeks prior to randomization
3. Palliative radiotherapy within 2 weeks, or radiotherapy for curative intent of target lesions within 8 weeks for chest and within 4 weeks for other areas prior to randomization
4. Major surgical procedure within 4 weeks prior to randomization
5. History of cardiac disease
6. Known symptomatic brain metastases
7. Need to breastfeed a child during or within 12 weeks of completing the study
8. Significant gastrointestinal disorder that could interfere with absorption of tivantinib and/or erlotinib
9. History of malignancy other than NSCLC
10. Known infection with HIV, active HBV or HCV
11. Clinically significant interstitial lung diseases detected by CT scan or prior history of such diseases
12. Psychiatric disease that could affect the informed consent process
13. Subjects who wish to have a child and who would not agree to use one or more contraceptive measures that are highly effective
14. Positive serum or urine pregnancy test in female subjects of childbearing potential
15. Any other significant co-morbid condition that, in opinion of the investigator/sub-investigator, would impair study participation or cooperation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-07; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression free survival
Objective response rate
  Each assessment will be determined based on RECIST criteria version 1.1 by investigator
Number of patients with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka, Japan

REFERENCES:
- [Derived] Yoshioka H, Azuma K, Yamamoto N, Takahashi T, Nishio M, Katakami N, Ahn MJ, Hirashima T, Maemondo M, Kim SW, Kurosaki M, Akinaga S, Park K, Tsai CM, Tamura T, Mitsudomi T, Nakagawa K. A randomized, double-blind, placebo-controlled, phase III trial of erlotinib with or without a c-Met inhibitor tivantinib (ARQ 197) in Asian patients with previously treated stage IIIB/IV nonsquamous nonsmall-cell lung cancer harboring wild-type epidermal growth factor receptor (ATTENTION study). Ann Oncol. 2015 Oct;26(10):2066-72. doi: 10.1093/annonc/mdv288. Epub 2015 Jul 7. PMID 26153496